CLINICAL TRIAL: NCT03869034
Title: Hepatic Arterial Infusion Chemotherapy Combined with PD-1 Inhibitor in Treating Potentially Resectable Locally Advanced Hepatocellular Carcinoma: a Prospective, Phase II Clinical Study
Brief Title: HAIC Combined with PD-1 Inhibitor in Potentially Resectable Locally Advanced HCC
Acronym: HAICPD1-HCC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Innovent Biologics, Inc. (Other)
Responsible Party: Principal Investigator, XU li, Clinical Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAICPD1-HCC
Record Dates: First submitted 2019-03-02; First posted 2019-03-11 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatic arterial Infusion Chemotherapy; PD-1 Inhibitor; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab

STUDY DESIGN:
Intervention Model Description: Patients enroll in this study will receive hepatic arterial infusion chemotherapy with FOLFOX regimen (FOLFOX-HAIC), or combined with Sintilimab PD-1 inhibitor.
Masking Description: None in this study will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A, Combination group (HAIC+PD-1) (Experimental): HAIC+PD-1
  Interventions: Combination Product: HAIC+PD1
- B, HAIC group (HAIC only) (Experimental): HAIC
  Interventions: Drug: HAIC

INTERVENTIONS:
Combination Product: HAIC+PD1 — Sintilimab ( 200mg Q3W iv D1)+FOLFOX-HAIC（oxaliplatin, 130 mg/m2 and leucovorin, 200 mg/m2, and fluorouracil, 400 mg/m2, bolus and 2400 mg/m2 over 46 hours Q3W D2 D3), maximally 8 cycles Multi-disciplinary consultation was organized to decide the chance of surgery and subsequent treatment per 2 treatment cycles. Patients who achieved partial response (PR) or minor response (MR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and were assessed as eligible for R0 resection go on to undergo surgical resection. After recovery from operation , sintilimab monotherapy was given per three weeks for maximally 16 doses. Patients who were ineligible for resection would continue to receive the combination therapy.
  Other Names: Sintilimab (IBI308); FOLFOX-HAIC
  Arms: A, Combination group (HAIC+PD-1)
Drug: HAIC — FOLFOX-HAIC: oxaliplatin, 130 mg/m2 and leucovorin, 200 mg/m2, and fluorouracil, 400 mg/m2, bolus and 2400 mg/m2 over 46 hours Q3W D2 D3, for maximally 8 cycles, and the safety parameters are reviewed before the start of each course of HAIC treatment. Patients who achieve partial response (PR) or minor response (MR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and are assessed as eligible for R0 resection go on to undergo surgical resection. No other anti-tumor therapies are allowed before PD or postoperative relapse is confirmed.
  Other Names: FOLFOX-HAIC
  Arms: B, HAIC group (HAIC only)

SUMMARY:
Hepatocellular carcinoma patients are mostly diagnosed at locally advanced stage. Nowadays, hepatic artery interventional therapy and/or systemic therapy are the main treatments options for these patients. Our previous study showed that compared to than conventional transcatheter arterial chemoembolization (TACE), hepatic arterial infusion chemotherapy (HAIC) has better objective response, better safety profile, and increased resection rates. The PD-1 inhibitors emerged in recent years have shown good momentum in the treatment of hepatocellular carcinoma. The single-drug treatment on advanced hepatocellular carcinoma has a tumor response rate of 17%, the disease control rate exceeds 60%, and the overall survival time exceeds 12 months. And it has good tolerance and less adverse events. In studies of other cancer, combined with traditional chemotherapy can further improve the efficacy of PD-1 inhibitors. Our study is a prospective phase II clinical study for patients with potentially resectable locally advanced hepatocellular carcinoma (tumor confined to the liver with invasion to branches of the portal vein or hepatic vein). Progressive survival (PFS) is the primary end point of study. The OS and overall survival rate, RFS, ORR, DCR, conversion rate, pathological response, and safety are the secondary endpoints. The efficacy and safety of HAIC combined with PD-1 inhibitor in the treatment of potentially resectable locally advanced hepatocellular carcinoma will be discussed.

DETAILED DESCRIPTION:
Sintilimab (IBI308) is a recombinant human IgG4 PD-1 monoclonal antibody. It has been proved in many preclinical and in vitro trials that the effect of blocking PD-1 pathway with Sintilimab on. The results of preclinical pharmacodynamics, animal pharmacokinetics and toxicology all indicated that Sintilimab has clear targets, reliable cell lines and drug stability. It has considerable characteristics and has shown good activity in various preclinical studies.

Hepatocellular carcinoma patients are mostly diagnosed in locally advanced stage, and hepatic artery interventional therapy and/or systemic therapy are the main treatments options for these patients. In recent years, some researchers have reported that chemotherapy plays a critical role in transcatheter arterial intervention (Shi et al. JNCI, 2012, 105: 59). Compared with transcatheter arterial chemoembolization (TACE), hepatic arterial infusion chemotherapy (HAIC) provides a more stable and long-lasting local control rate, which promised better outcomes. However, the effectiveness of HAIC varies greatly depending on the chemotherapy drug used, with an efficiency ranging from 7-81% and OS ranging from 6-15.9 months.

The single-drug treatment of PD-1 inhibitor in advanced hepatocellular carcinoma has a tumor response rate of 17%, the disease control rate exceeds 60%, and the overall survival time exceeds 12 months. And it has good tolerance and less adverse events. In studies in other cancers, combined with traditional chemotherapy can further improve the efficacy of PD-1 inhibitors.

Our study is a prospective phase II clinical study for patients with potentially resectable locally advanced hepatocellular carcinoma (tumor confined to the liver with invasion to branches of the portal vein or hepatic vein). Progressive survival (PFS) based on RECIST 1.1 is the primary end point of the present study. The OS and overall survival rate, RFS, ORR, DCR, conversion rate, pathological response, and safety are the secondary endpoints. The exploratory endpoints included the research on biomarkers. The efficacy and safety of HAIC combined with PD-1 inhibitor in the treatment of potentially resectable locally advanced hepatocellular carcinoma will be discussed.

Radiological assessments are performed every two cycles over the course of treatment, then every 3 months within the first two years following the completion of treatment and every 6 months thereafter, until PD were recorded. All subjects are followed until death or lost to follow up. The recurrence, metastasis sites, detection methods, adjuvant treatment and accurate survival time were recorded in detail.

Due to the lack of historical data and expected effect size for this population, the sample size of this pilot study is arbitrarily set at 40, including two intervention arms. Arm A will included 30 patients who receive HAIC combined with sintilimab. Arm B will included 10 patients who receive only HAIC. The patients are assigned to any group according to their willing.

The Kaplan-Meier method was used to estimate progression-free survival and overall survival; the Log-rank method was used for single factor analysis; the Cox model was analyzed by multivariate analysis. All the statistical tests were two-sided, and P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 years and 70 years.
2. Hepatocellular carcinoma: patients need to be diagnosed as hepatocellular carcinoma (HCC) histologically before treatment.
3. Never received any anti-cancer treatment in the past.
4. potentially resectable Locally advanced HCC: with at least one measurable lesion (RECIST 1.1), and tumor(s) confined to the left or right hemi-liver, with macroscopic invasion to branch of the portal vein and/or hepatic vein.
5. No extrahepatic metastases.
6. No contraindications for the treatment of HAIC and PD-1 inhibitors.
7. KPS≥90.
8. Liver function: Child-Pugh class A.
9. The expected survival of the patient is more than 6 months.
10. Adequate hematological and organ function.
11. The following conditions are met:

    Platelet≥75×10^9/L; White blood cell≥3.0×10^9/L; Hemoglobin≥90 g/L; Serum creatinine≤1.5 × upper limit of normal (ULN); PT≤3 second extension; total bilirubin ≤1.5 x ULN； AST and ALT ≤2.5 x ULN.
12. Agree to accept postoperative follow-up required by the design of this study.
13. Patients must have the ability to understand and voluntarily sign the informed consent, and must sign an informed consent before starting any specific procedure for the study.

Exclusion Criteria:

1. In combined with severe heart, lung, kidney or other important organ dysfunction, or combined with serious infection or other serious associated diseases, that cannot tolerate treatment (> CTCAE Version 4.03 adverse events of grade 2).
2. With uncontrolled hepatitis B (HBV-DNA>2000 IU/ml and elevated ALT).
3. Multi-nodules hepatocellular carcinoma beyond hemi-hepatic range.
4. Patients with tumor thrombus reaches or exceeds the portal vein.
5. History of other malignancies.
6. History of allergic reactions to related drugs.
7. History of organ transplantation.
8. Pregnant women, nursing mothers.
9. Patients have other factors that may interfere with patient enrollment and assessment results.
10. Refuse follow-up as required by this study protocol and refuse to sign informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) assessed by RECIST 1.1 | From date of the first treatment until the date of progression or death from any cause, whichever occurs first, assessed up to 96 months
  The duration from treatment initiation to disease progression or death from any cause in patients who did not undergo surgery, or to the date of postoperative relapse or death from any cause in patients who had received surgery, whichever occurs first. The baseline of the tumor before the initial treatment was used as a reference, and the assessments are performed according to the RECIST 1.1 criteria based on the imaging test (enhanced CT or MRI).

SECONDARY OUTCOMES:
Overall survival (OS) | From date of the first treatment until the date of death from any cause, assessed up to 96 months
  The time between the first HAIC +PD1 treatment and death from any cause.
1-, 2- and 3-year Overall Survival (OS) rate | From date of the first treatment until the date of death from any cause, assessed up to 96 months
  The percentage of patients who were still alive at the 1-, 2-, and 3-year time point since the first cycle of treatment. The end point of observation is death due to tumor.
Safety: the percentage of participants with treatment-related adverse events as assessed by CTCAE v4.03 | From date of the first treamtment until 100 days after the last treatment.
  adverse events will be assessed and reported according to NCI CTC AE v4.03.
Pathological Response: pathological complete response (pCR) and major pathological response (MPR: >90% of tumor necrosis) | Through study completion, an average of 1 year.
  According to post-operative pathology, the proportion of tumor necrosis, viable. tumor cells, and tumor infiltrating lymphocytes indicated by surgical resected specimens.
Objective Response Rate (ORR) assessed by RECIST 1.1 | Through study completion, an average of 3 year.
  The proportion of complete response or partial response as optimal response among all treated patients.
Disease Control Rate (DCR) | Through study completion, an average of 3 year.
  The proportion of complete response, partial response or stable disease as optimal response assessed by RECIST 1.1 among all treated patients.
Conversion rate | Through study completion, an average of 1 year.
  The proportion of patients who received surgical resection among all treated patients.
Recurrence-free survival (RFS) | From date of the surgery until the date of first recurrence/metastasis after resection or death from any cause, assessed up to 96 months
  The time between surgery and first recurrence/metastasis after resection or death from any cause, whichever occurs first.

OTHER OUTCOMES:
Biomarkers of treatment response by single-cell RNA sequencing | From date of first dose until the date of first documented progression, assessed up to 96 months
  To find biomarkers of treatment response by investigating the variation of tumor and immune cells before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Min-shan Chen, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be openly available in Research Data Deposit at https://www.researchdata.org.cn/default.aspx, after publication.
Supporting Information: CSR
Time Frame: since publication
Access Criteria: open
URL: http://www.researchdata.org.cn

REFERENCES:
- [Background] Lyu N, Kong Y, Mu L, Lin Y, Li J, Liu Y, Zhang Z, Zheng L, Deng H, Li S, Xie Q, Guo R, Shi M, Xu L, Cai X, Wu P, Zhao M. Hepatic arterial infusion of oxaliplatin plus fluorouracil/leucovorin vs. sorafenib for advanced hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):60-69. doi: 10.1016/j.jhep.2018.02.008. Epub 2018 Feb 20. PMID 29471013
- [Background] Lyu N, Lin Y, Kong Y, Zhang Z, Liu L, Zheng L, Mu L, Wang J, Li X, Pan T, Xie Q, Liu Y, Lin A, Wu P, Zhao M. FOXAI: a phase II trial evaluating the efficacy and safety of hepatic arterial infusion of oxaliplatin plus fluorouracil/leucovorin for advanced hepatocellular carcinoma. Gut. 2018 Feb;67(2):395-396. doi: 10.1136/gutjnl-2017-314138. Epub 2017 Jun 7. No abstract available. PMID 28592441
- [Background] He MK, Le Y, Li QJ, Yu ZS, Li SH, Wei W, Guo RP, Shi M. Hepatic artery infusion chemotherapy using mFOLFOX versus transarterial chemoembolization for massive unresectable hepatocellular carcinoma: a prospective non-randomized study. Chin J Cancer. 2017 Oct 23;36(1):83. doi: 10.1186/s40880-017-0251-2. PMID 29061175
- [Derived] Pan Y, Wang X, Peng C, Zhao J, Lu S, Zhang C, Wang J, Fu Y, Zhou Z, Chen M, Zhang Y, Xu L. Hepatic arterial infusion chemotherapy plus sintilimab as conversion therapy for locally advanced hepatocellular carcinoma: a single-center phase II trial. Int J Surg. 2026 Jan 13. doi: 10.1097/JS9.0000000000004692. Online ahead of print. PMID 41537370